CLINICAL TRIAL: NCT03670836
Title: Dilapan vs Misoprostol for Cervical Ripening [COMRED - Comparison of Misoprostol Ripening Efficacy With Dilapan]
Brief Title: Comparison of Misoprostol Ripening Efficacy With Dilapan
Acronym: COMRED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Medicem International CR s.r.o. (Industry)
Responsible Party: Principal Investigator, Rachana Gavara, Assistant Professor of Obstetrics and Gynecology at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAR8566
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Labor Onset and Length Abnormalities; Induced; Birth
Keywords: Misoprostol; Dilapan; Induction of labor; Aquacryl hydrogel
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dilapan group (Experimental): Patients who are randomized to receive Dilapan, will have 3-5 rods of Dilapan-S® inserted in their cervix by the supervising provider, under aseptic precautions with a speculum exam, either digitally or using a sponge forceps, as per manufacturer's recommendations. The Bishop score at the time of eligibility assessment and number of rods inserted will be recorded. Dilapan will be left in cervix for 12 hours. Patients will be allowed to ambulate, shower and have light meals as long as they meet the criteria based on institutional guidelines for intermittent fetal heart monitoring. "Nothing per vagina" including douching and no bathing is allowed.
  Interventions: Device: Dilapan
- Misoprostol group (Experimental): Patients who are randomized to Misoprostol group, after the baseline assessment and a reassuring cardiotocograms (CTG) monitoring for 20 minutes to a maximum of 6 doses. All subjects will have continuous fetal monitoring. A dose will be held if patient is noted to have uterine tachysystole, hyperstimulation, fetal heart tracing abnormalities or 3 or more painful uterine contractions over a period of 10 minutes (indicating onset of labor). Administration of Misoprostol will be done by the nurse assigned to the patient.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Device: Dilapan — Dilapan-S® is a mechanical method for cervical ripening using rods made of a patented hydrogel Aquacryl, it is marketed in form of rods of 3 and 4 mm diameter. It is FDA approved for cervical ripening.
  Other Names: Aquacryl Hydrogel
  Arms: Dilapan group
Drug: Misoprostol — 25mcg of Misoprostol will be administered orally every 2 hours (maximum of 6 doses)
  Misoprostol is a prostaglandin E1 analog approved for treatment and prevention of gastric ulcers. The use of Misoprostol appears to be safe and effective for induction of labor when used in low dose.
  Other Names: Cytotec
  Arms: Misoprostol group

SUMMARY:
The purpose of this study is to find out if Dilapan works as well as Misoprostol for preparing the mouth of the uterus (cervix) for inducing labor in women who need to undergo this procedure. The primary objective is to assess the efficacy of Dilapan for cervical ripening compared to Misoprostol in women undergoing Induction of labor (IOL) at or more than 37 weeks gestation.

DETAILED DESCRIPTION:
In developed nations 25 % of pregnant women undergo labor induction for various indications. Likelihood of vaginal delivery depends on the degree of ripeness of cervix. Majority of women undergoing induction of labor are candidates for cervical ripening. Dilapan is an osmotic hygroscopic dilator of cervix commonly used for cervical preparation for mid trimester abortions. It has been proven safe for use for induction of Labor (IOL) at term. Misoprostol is a synthetic prostaglandin E1 analogue, widely used for cervical ripening and IOL in United States and is considered as standard of care.

This is a non-inferiority, unblinded randomized, controlled trial where 322 eligible participants undergoing IOL at >37 weeks gestation and admitted to labor and delivery unit will be enrolled and randomly assigned in a ratio 1:1 to either receive Dilapan or Misoprostol for cervical ripening.

After randomization all participants will undergo assessment as per standard of care. Participants will have either 1-5 Dilapan rods inserted into their cervix by the providers or receive 25 mcg of misoprostol orally every 2 hours to a maximum of 6 doses over 12 hours. Participants will be evaluated for artificial rupture of membranes and initiation of oxytocin for inducing uterine contraction. A diagnosis of failed IOL will be made if patient does not go into active labor within 24 hours after initiation of Oxytocin and Artificial Rupture Of Membranes (AROM). Intrapartum management will be according to institutional guidelines. All participants will be followed up and contacted by phone 2 weeks after discharge regarding their experience with the method of induction.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing labor induction with a gestation of ≥37 weeks (based on a sure last menstrual period and an ultrasound done before 22 0/7 weeks)
2. Live fetus with in cephalic presentation
3. Singleton pregnancy
4. Able to provide informed consent for participation in the study

Exclusion Criteria:

1. Contraindication for vaginal delivery
2. Age less than 18 years
3. Prior uterine scar from a cesarean section or myomectomy
4. Patients who have HELLP syndrome or eclampsia
5. Active genital herpes at the time of labor induction
6. Complex medical problems that may require assistance with second stage of labor
7. Bishop score ≥ 6
8. Major fetal congenital anomalies (as assessed by investigator)
9. Premature rupture of membranes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachana Gavara, MD, Principal Investigator — rg2460@cumc.columbia.edu
Locations (2):
- United States (2):
  - New York Presbyterian - Allen Hospital, New York, New York
  - University of Texas, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Gavara R, Saad AF, Wapner RJ, Saade G, Fu A, Barrow R, Nalgonda S, Bousleiman S, Almonte C, Alnafisee S, Holman A, Burgansky A, Heikkila P. Cervical Ripening Efficacy of Synthetic Osmotic Cervical Dilator Compared With Oral Misoprostol at Term: A Randomized Controlled Trial. Obstet Gynecol. 2022 Jun 1;139(6):1083-1091. doi: 10.1097/AOG.0000000000004799. Epub 2022 May 2. PMID 35675605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1755 women presenting for Induction of labor to labor and delivery units were screened for eligibility at Columbia University Medical Center and UTMB Texas. 307 were enrolled and randomized, 154 to Dilapan and 153 to Oral Misoprostol group.
Pre-assignment Details: A total of 306 participants were needed , 153 in each group, to evaluate the primary outcome with 85% power to confirm the noninferiority with one sided confidence level of 97.5%
Groups:
- Misoprostol Group- 153: Patients who are randomized to Misoprostol group, after the baseline assessment and a reassuring cardiotocograms (CTG) monitoring for 20 minutes to a maximum of 6 doses. All subjects will have continuous fetal monitoring. A dose will be held if patient is noted to have uterine tachysystole, hyperstimulation, fetal heart tracing abnormalities or 3 or more painful uterine contractions over a period of 10 minutes (indicating onset of labor). Administration of Misoprostol will be done by the nurse assigned to the patient.
  Misoprostol: 25mcg of Misoprostol will be administered orally every 2 hours (maximum of 6 doses)
  Misoprostol is a prostaglandin E1 analog approved for treatment and prevention of gastric ulcers. The use of Misoprostol appears to be safe and effective for induction of labor when used in low dose.
- Dilapan Group 154: Patients who are randomized to receive Dilapan, will have 3-5 rods of Dilapan-S® inserted in their cervix by the supervising provider, under aseptic precautions with a speculum exam, either digitally or using a sponge forceps, as per manufacturer's recommendations. The Bishop score at the time of eligibility assessment and number of rods inserted will be recorded. Dilapan will be left in cervix for 12 hours. Patients will be allowed to ambulate, shower and have light meals as long as they meet the criteria based on institutional guidelines for intermittent fetal heart monitoring. "Nothing per vagina" including douching and no bathing is allowed.
  Dilapan: Dilapan-S® is a mechanical method for cervical ripening using rods made of a patented hydrogel Aquacryl, it is marketed in form of rods of 3 and 4 mm diameter. It is FDA approved for cervical ripening.
Period: Intent-to-treat Population (ITT)
Arm/Group | Misoprostol Group- 153 | Dilapan Group 154
Started (Enrollment period was from Nov 2018) | 153 | 154
Completed (Jan 31st 2021) | 152 | 151
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Period: Per Protocol Population (PP)
Arm/Group | Misoprostol Group- 153 | Dilapan Group 154
Started (Patients randomized to each group) | 152 | 151
Completed (Completed the protocol) | 138 | 134
Not Completed | 14 | 17
Not completed — Physician Decision | 9 | 10
Not completed — Physician Decision | 4 | 6
Not completed — Incorrect stratification / inability to insert Dilapan | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics were analyzed in the intent to treat population
Groups:
- Misoprostol Group: Patients who are randomized to Misoprostol group, after the baseline assessment and a reassuring cardiotocograms (CTG) monitoring for 20 minutes to a maximum of 6 doses. All subjects will have continuous fetal monitoring. A dose will be held if patient is noted to have uterine tachysystole, hyperstimulation, fetal heart tracing abnormalities or 3 or more painful uterine contractions over a period of 10 minutes (indicating onset of labor). Administration of Misoprostol will be done by the nurse assigned to the patient.
  Misoprostol: 25mcg of Misoprostol will be administered orally every 2 hours (maximum of 6 doses)
  Misoprostol is a prostaglandin E1 analog approved for treatment and prevention of gastric ulcers. The use of Misoprostol appears to be safe and effective for induction of labor when used in low dose.
- Total: Total of all reporting groups
Arm/Group | Dilapan Group | Misoprostol Group | Total
Number analyzed (Participants) | 151 | 152 | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.2 (5.94) | 27.7 (5.9) | 27.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 152 | 303
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gestational age at randomization < 39 weeks [Count of Participants; unit: Participants]
  Gestational age ≤ 39 weeks | 57 | 55 | 112
  Gestational age > 39 weeks | 94 | 97 | 191
Parity at randomization- Nulliparous/ multiparous [Count of Participants; unit: Participants]
  Nulliparous | 81 | 81 | 162
  Multiparous | 70 | 71 | 141
BMI at randomization [Mean (Standard Deviation); unit: kg/m^2] | 33.1 (5.02) | 33.1 (4.83) | 33.1 (5.9)
GBS positive status [Count of Participants; unit: Participants] | 60 | 52 | 112
Indication for induction - Diabetes [Count of Participants; unit: Participants] | 15 | 7 | 22
Hypertensive disorders of pregnancy [Count of Participants; unit: Participants] | 14 | 20 | 34
Post term pregnancy [Count of Participants; unit: Participants] | 47 | 40 | 87
Fetal growth restriction [Count of Participants; unit: Participants] | 9 | 6 | 15
Oligohydramnios [Count of Participants; unit: Participants] | 14 | 22 | 36
Cholestasis [Count of Participants; unit: Participants] | 1 | 2 | 3
Elective induction [Count of Participants; unit: Participants] — Number of participants who underwent elective induced labor
  Participants | 37 | 32 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Achieving Vaginal Delivery Within 36 Hours After Initiation of Cervical Ripening in ITT Population
Description: This is to measure the efficacy of either Dilapan or Misoprostol for cervical ripening.
  Intent-to-treat Population (ITT) includes all patients that were randomized into the study. ITT participants will be analyzed in accordance with their randomized study treatment (i.e. in the treatment group they were originally allocated, regardless of treatment actually received). ITT will be used for evaluation of the baseline characteristics and as the primary population for efficacy assessments.
Time Frame: Up to 36 hours after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 93 | 90

2. Primary Outcome: Number of Women Achieving Vaginal Delivery Within 36 Hours After Initiation of Cervical Ripening in PP Population
Description: This is to measure the efficacy of either Dilapan or Misoprostol for cervical ripening.
Time Frame: Up to 36 hours after intervention
Population: The Per Protocol (PP) population is a subset of ITT population. PP population is comprised of participants who completed the treatment originally allocated with complete adherence to the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 134 | 138
Participants | 86 | 86

3. Secondary Outcome: Change in Bishop Score
Description: The Bishop Score (also known as Pelvic Score) is the most commonly used method to rate the readiness of the cervix for induction of labor. The Bishop Score gives points to 5 measurements of the pelvic examination dilation, effacement of the cervix, station of the fetus, consistency of the cervix, and position of the cervix. It ranges from 0 to 13. Higher score is associated with increased likelihood of vaginal delivery.
Time Frame: Baseline and 12 hours after intervention
Population: Intent to treat population
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
score on a scale | 2 [0 to 11] | 3 [0 to 11]

4. Secondary Outcome: Percentage of Women Delivering Vaginally in 24 Hours After the Initiation of Intervention
Description: This is to measure the efficacy of either Dilapan or Misoprostol for cervical ripening
Time Frame: Up to 24 hours after intervention
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 62 | 58

5. Secondary Outcome: Overall Vaginal Delivery Rate
Description: This is to measure the efficacy of either Dilapan or Misoprostol for cervical ripening
Time Frame: Approximately up to 48 hours
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 104 | 104

6. Secondary Outcome: Number of Participants With Cesarean Deliveries
Description: This is to measure the efficacy of either Dilapan or Misoprostol for cervical ripening
Time Frame: Start of cervical ripening to delivery, up to 36 hours
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 41 | 42

7. Secondary Outcome: Total Length of Hospital Stay
Description: This is to measure the cost-effectiveness of either Dilapan or Misoprostol for cervical ripening. Length will be measured in number of days from hospital admission until discharge.
Time Frame: Up to 4 days
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
hours | 80.5 (21.8) | 84.0 (22.6)

8. Secondary Outcome: Percentage of Women Who Developed Chorioamnionitis
Description: This is to measure the safety of either Dilapan or Misoprostol for cervical ripening
Time Frame: From delivery until two weeks after discharge (approximately up to 3 weeks)
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 12 | 10

9. Secondary Outcome: Percentage of Women Who Developed Postpartum Hemorrhage
Description: This is to measure the safety of either Dilapan or Misoprostol for cervical ripening, postpartum hemorrhage is defined as estimated blood loss (EBL) > 1000cc and/or drop in Hematocrit (HCT) by 10 points.
Time Frame: From delivery until two weeks after discharge (approximately up to 3 weeks)
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 1 | 3

10. Secondary Outcome: Percentage of Newborns With Apgar Score <7 at 5 Min
Description: This is to measure the safety of either Dilapan or Misoprostol for cervical ripening by studying the effect on newborns
Time Frame: 5 minutes following birth
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 0 | 1

11. Secondary Outcome: Percentage of Newborns With Cord Arterial Blood Potential Hydrogen (pH) < 7.1
Description: This is to measure the safety of either Dilapan or Misoprostol for cervical ripening by studying the effect on newborns
Time Frame: From birth until two weeks after birth
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 0 | 4

12. Secondary Outcome: Percentage of Newborns With Neonatal Intensive Care Unit (NICU) Admission Within 14 Days After Study Intervention
Description: This is to measure the safety of either Dilapan or Misoprostol for cervical ripening by studying the effect on newborns
Time Frame: From birth until two weeks after birth
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 9 | 8

13. Secondary Outcome: Percentage of Newborns With Antibiotic Use Within 14 Days After Study Intervention
Description: This is to measure the safety of either Dilapan or Misoprostol for cervical ripening by studying the effect on newborns
Time Frame: From birth until two weeks after birth
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Dilapan Group | Misoprostol Group
Number analyzed (Participants) | 151 | 152
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: Data was collected from the time of randomization to 2 weeks after delivery for the enrolled subjects and their neonates .
Description: A serious event is defined a new condition that develops during the course of study and will require significantly higher level of care like transfer to ICU for blood transfusion of multiple units .
Arm/Group | Dilapan Group | Misoprostol Group
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/152
Serious Adverse Events (participants affected / at risk) | 1/151 | 3/152
Other Adverse Events (participants affected / at risk) | 39/151 | 81/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dilapan Group (N=151) | Misoprostol Group (N=152)
postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) — Blood loss of more than 1000cc immediately after delivery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dilapan Group (N=151) | Misoprostol Group (N=152)
uterine tachysystole (Pregnancy, puerperium and perinatal conditions) | 35 (35) | 70 (70) — Too frequent uterine contractions during labor induction
uterine tachy systole with abnormal fetal heart tracing (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT03670836/Prot_002.pdf
  • Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT03670836/SAP_001.pdf